CLINICAL TRIAL: NCT07125729
Title: ctDNA Testing in Resectable Stage II-IV Colorectal Cancer Patients: A Head-to-Head Performance Comparison
Brief Title: Minimal Residual Disease Testing for the Early Detection of Cancer Recurrence in Resectable Stage II-IV Colorectal Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 24372; NCI-2025-05428 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24372 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-08-10; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Resectable Colorectal Carcinoma; Stage II Colorectal Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Specimen Handling; Cell-Free Nucleic Acids; Circulating Tumor DNA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening (Haystack MRD, Signatera) (Experimental): Patients undergo archival tissue and blood sample collection and Haystack MRD and Signatera ctDNA/cfDNA testing prior SOC surgical resection. Patients then undergo blood sample collection and Haystack MRD and Signatera ctDNA/cfDNA testing 3-10 weeks after surgery, every 3 months for 2 years post-surgery, and then every 6 months for years 3-5 post-surgery in the absence of disease progression.
  Interventions: Procedure: Biospecimen Collection; Other: cfDNA or ctDNA Measurement; Other: Electronic Health Record Review

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo archival tissue and/or blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: cfDNA or ctDNA Measurement — Undergo Haystack MRD and Signatera ctDNA/cfDNA testing
  Other Names: Cell-Free DNA/Circulating Tumor DNA Measurement; cfDNA/ctdDNA Measurement; cfDNA/ctDNA; cfDNA/ctDNA Measurement; Circulating Cell-Free DNA/Circulating Tumor-Derived DNA Measurement
Other: Electronic Health Record Review — Ancillary studies

SUMMARY:
This clinical trial compares minimal residual disease (MRD) testing with the Haystack blood test (assay) to the Signatera® assay for the early detection of the cancer returning (cancer recurrence) in patients with stage II-IV colorectal cancer (CRC) that can be removed by surgery (resectable). MRD testing looks for evidence of remaining tumor following treatment that is only apparent using highly sensitive techniques. There are few effective tools available outside of imaging to identify CRC patients with MRD who may be at the highest risk for cancer recurrence after surgery. Early detection of CRC recurrence after surgery is important, as it may increase the chance of curative (ability to cure) outcomes for patients with cancer recurrence. Currently, the Signatera assay is used to monitor whether CRC recurs after surgery, however it is not a very sensitive test. Early work with the Haystack assay suggests it may be more sensitive than the Signatera assay, which may be more effective for the early detection of cancer recurrence in patients with resectable stage II-IV CRC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the clinical performance of the Haystack MRD test and the Signatera® test in patients with stage II-IV CRC patients treated with curative intent surgery with or without adjuvant therapy.

SECONDARY OBJECTIVE:

I. To calculate the lead time (months) of recurrence detection by the Haystack MRD test in curatively resected colorectal cancer patients to 1) radiological recurrence time 2) Signatera® test positivity.

EXPLORATORY OBJECTIVE:

I. To explore the performance of up to two cancer detection assays (BestSEEK and enACT) in development by Dr. Tomasetti at City of Hope - Translational Genomics Research Institute (TGen) and City of Hope.

OUTLINE:

Patients undergo archival tissue and blood sample collection and Haystack MRD and Signatera circulating tumor deoxyribonucleic acid (ctDNA)/cell-free deoxyribonucleic acid (cfDNA) testing prior to standard of care (SOC) surgical resection. Patients then undergo blood sample collection and Haystack MRD and Signatera ctDNA/cfDNA testing 3-10 weeks after surgery, every 3 months for 2 years post-surgery, and then every 6 months for years 3-5 post-surgery in the absence of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Documented written informed consent of the participant
* Age: ≥ 18 years
* Diagnosis of stage II, III or IV colorectal cancer (any gender) if enrolled post-operatively. If a treatment naïve patient is enrolled pre-operatively and determined to be pathological stage I, the patient will be replaced
* Patient who are to undergo a curative intent surgery or have undergone a curative resection and are presenting for surveillance
* Patient identified as an appropriate candidate for Signatera® testing as a standard of care MRD surveillance assay
* Patient willingness to continue Signatera® assay every 3 months for 2 years in the first 2 years after resection and every 6 months for years 3, 4, 5 after resection, as performed by standard of care testing. In addition, the patients should be willing to provide blood samples for Haystack MRD testing at the same intervals of Signatera®, along with willingness to allow access to archival tissue to allow for Haystack MRD assay personalization. Surveillance with ctDNA should be initiated between 3 to 10 weeks from surgery
* Adequate availability of archival tissue or anticipated pathological viable tissue. All untreated primary resection would be expected to have adequate tissue. Patients with resected metastatic disease should have either previously resected primary that is amenable for tumor informed MRD testing or should have adequate archival metastasectomy samples
* Patients with total neoadjuvant therapy (TNT) for rectal cancer and complete clinical response with plans of watchful waiting may also be enrolled as long as there is adequate tissue from prior endoscopic biopsies to allow for Signatera® and Haystack MRD assays

Exclusion Criteria:

* Inability to safely provide sequential blood samples
* Clinical evidence of unresected metastatic disease
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-07-12 (Actual); Primary Completion 2028-01-09 (Estimated); Study Completion 2028-01-09 (Estimated)

PRIMARY OUTCOMES:
Minimal residual disease (MRD) rate with Haystack and Signatera® | Up to 5 years
  Will assess the MRD rate with Haystack (positive circulating tumor deoxyribonucleic acid [+ctDNA] and negative imaging) versus MRD rate with Signatera (+ctDNA and negative imaging). Sensitivity (i.e., true positive rate - proportion of patients who recur that are found to be MRD positive), specificity (i.e., true negative rate - proportion of patients who do NOT recur that are found to be MRD negative), positive predictive value (i.e., proportion of positive tests which are true positives) and negative predictive value (proportion of negative tests which are true negatives) of the Haystack test and of the Signatera test for predicting disease recurrence will be calculated and summarized at various times of testing.

SECONDARY OUTCOMES:
Time interval of detection of disease recurrence by Haystack test, radiological imaging, and Signatera test | Up to 5 years
  The time interval between recurrence detection by the Haystack MRD test compared to radiological imaging assessment and Signatera test will be calculated as the time interval between the detection of disease recurrence by each of the methods (Haystack test, radiological imaging, Signatera test). Lead-time will be estimated by means of appropriate formulas and Monte Carlo simulation. Pairwise comparisons of detection times will be performed using the log-rank test. Cox proportional hazards model will be used to estimate the hazard ratios and 95% confidence intervals for each detection method.
Level of association of circulating tumor deoxyribonucleic acid (ctDNA) result and status of recurrence and non-recurrence | Up to 5 years
  Logistic regression model will be used to estimate the level of association of ctDNA result and the status of recurrence and non- recurrence in patients with resectable stage II-IV colorectal cancer. Multivariable models adjusting for relevant clinical variables will be evaluated to assess the importance of these prognostic factors and support the robustness of ctDNA findings.

CONTACTS AND LOCATIONS:
Overall Officials: Marwan G Fakih, Principal Investigator — City of Hope Medical Center
Locations (13):
- United States (13):
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - City of Hope Corona, Corona, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope Seacliff, Huntington Beach, California
  - City of Hope at Irvine Lennar, Irvine, California
  - City of Hope Antelope Valley, Lancaster, California
  - City of Hope at Long Beach Elm, Long Beach, California
  - City of Hope at Newport Beach Fashion Island, Newport Beach, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope South Bay, Torrance, California
  - City of Hope Upland, Upland, California
  - City of Hope Atlanta Cancer Center, Newnan, Georgia
  - City of Hope at Chicago, Zion, Illinois